CLINICAL TRIAL: NCT03471130
Title: A Phase I, Randomised, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Effect of MT-8554 at Two Dose Levels, MT-8554 Low Dose and MT-8554 High Dose, on the QT/QTc Interval in Healthy Adult Subjects
Brief Title: Definitive QT Study With MT-8554
Acronym: MT-8554 DQT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MT-8554-E08; 2017-004138-27 (EudraCT Number)
Record Dates: First submitted 2018-02-28; First posted 2018-03-20 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Intervention Model Description: Double blind, placebo controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose MT-8554 or placebo to match (Experimental): Low dose MT-8554
  Interventions: Drug: MT-8554 Low dose; Drug: Placebo
- High dose MT-8554 or placebo to match (Experimental): High dose MT-8554
  Interventions: Drug: MT-8554 High dose; Drug: Placebo

INTERVENTIONS:
Drug: MT-8554 Low dose — Oral, 7 days
  Arms: Low dose MT-8554 or placebo to match
Drug: MT-8554 High dose — Oral, 7 days
  Arms: High dose MT-8554 or placebo to match
Drug: Placebo — Oral, 7 days

SUMMARY:
This is a study to definitively assess the effects of MT 8554, adjusted for placebo, on the change of the QT interval corrected for heart rate (HR) using the Fridericia formula (QTcF) from Baseline in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

* 1. Provide written informed consent to participate in this study.
* 2. Healthy and free from clinically significant illness or disease as determined by medical history, physical examination (PE), laboratory, and other tests at Screening and Admission.
* 3. Male and female subjects, aged 18 to 55 years (inclusive) at Screening.
* 4. A body weight of ≥60 kg male and ≥50 kg female and a body mass index ranging from 18 to 30 kg/m2 (inclusive) at Screening.
* 5. Subjects and partners agree to use contraception throughout the study as detailed in the protocol.
* 6. In the Investigator's opinion, subject is able to understand the nature of the study and any risks involved in participation, and willing to cooperate and comply with the protocol restrictions and requirements.

Exclusion Criteria:

* 1. Subjects with PR >240 ms, QRS ≥120 ms or corrected QT interval (QTc) by Fridericia's correction >450 ms for males and >470 ms for females on the Screening ECG, or any clinically significant ECG abnormality, in the opinion of the Investigator.
* 2. Subjects who have a history of cardiac disease or arrhythmias that can cause QTc prolongation.
* 3. Family history of long or short QT syndrome, hypokalaemia, syncope, or Torsades de Pointes.
* 4. Clinically significant (in the opinion of the Investigator) endocrine, thyroid, hepatic (including Gilbert's syndrome), respiratory, gastrointestinal (GI), renal (including estimated glomerular filtration rate <90 mL/min), cardiovascular disease, or history (within the last 2 years) of any significant psychiatric/psychotic illness disorder (including anxiety, depression and reactive depression).
* 5. Clinically relevant abnormal medical history, physical findings, or laboratory values at Screening or Day -1 that could interfere with the objectives of the study or the safety of the subject, as judged by the Investigator.
* 6. Previously having received MT-8554.
* 7. Participation in more than 3 clinical studies involving administration of an IMP in the previous year, or any study within 12 weeks (or if relevant, 5 half-lives, whichever is longer) prior to the first dose.
* 8. Presence or history of severe adverse reaction or allergy to any medicinal product that is of clinical significance.
* 9. Subjects who have received any prescribed systemic or topical medication within 14 days (or if relevant, 5 half-lives; whichever is longer) prior to the first dose of IMP unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with the study procedures or compromise safety. Subjects who have received slow release medicinal formulations considered to still be active within 14 days (or if relevant, 5 half-lives; whichever is longer) prior to the first dose administration will also be excluded unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with the study procedures or compromise subject safety.
* 10. Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days (or, if relevant, five half-lives; whichever is longer) prior to the first dose of IMP unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with the study procedures or compromise safety. Occasional use of paracetamol (acetaminophen) for mild analgesia is permitted.
* 11. Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days (or if relevant, 5 half lives; whichever is longer) prior to the first dose of IMP unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with the study procedures or compromise safety.
* 12. Subjects with aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≥1.5×upper limit of normal (ULN) or total bilirubin or creatine kinase above the reference range at Screening or Day -1.
* 13. Blood pressure (BP, supine) at Screening or Day -1 outside the range 90 to 140 mmHg (systolic) or 50 to 90 mmHg (diastolic); and pulse rate outside the range of 40 to 100 beats per minute (bpm), confirmed by repeat assessment. Evidence of postural hypotension defined as a decrease of >20 mmHg in systolic bp or >10 mmHg in diastolic bp between the supine and standing position, confirmed by repeat assessment.
* 14. Tympanic body temperature at Day -1 that is outside the local reference range, confirmed by repeat assessment.
* 15. Subjects who are pregnant (positive pregnancy test at Screening or Day -1) or lactating.
* 16. Presence or history of lactose intolerance.
* 17. Excessive consumption of food or drink containing caffeine, including coffee, tea, cola, energy drinks or chocolates (>5 cups of coffee or equivalent per day).
* 18. Presence or history of drug abuse (as defined by Diagnostic and Statistical Manual of Mental Disorders [DSM-V] criteria), or a positive urine test for drugs of abuse at Screening or Day 1.
* 19. Presence or history (in the last 2 years) of alcohol abuse, or intake of more than 28 units/224 g of alcohol weekly (for men) or 21 units/168 g of alcohol weekly (for women) or a positive breath test for alcohol at Screening or Day -1. One unit/8 g is equivalent to a half-pint (280 mL) of beer, 1 measure (25 mL) of spirits, or 1 glass (125 mL) of wine.
* 20. Subjects who use tobacco or nicotine-containing products (cigarettes, snuff, chewing tobacco, cigars, pipes, e-cigarettes or nicotine replacement products) within 3 months prior to dosing, or positive urine cotinine test at Screening or Day -1.
* 21. Test positive for hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody, or human immunodeficiency virus (HIV) 1 & HIV 2 antibodies at Screening.
* 22. Donate ≥1 units of blood (450 mL) in the 3 months prior to Screening, plasma in the 7 days prior to Screening, platelets in the 6 weeks prior to Screening, or intention to donate blood within 3 months after the last scheduled visit.
* 23. Consumption of food or drink containing Seville oranges, cranberry, liquorice or grapefruit from 7 days prior to Day -1.
* 24. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs; or which may jeopardise the subject in case or participation in the study. The Investigator should be guided by evidence of any of the following histories:

  1. Inflammatory bowel syndrome, gastritis, ulcers, GI or rectal bleeding
  2. Major GI surgery such as gastrectomy, gastroenterostomy, or bowel resection
  3. Clinical evidence of pancreatic injury or pancreatitis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QTcF with placebo adjustment | Days 1 & 7

SECONDARY OUTCOMES:
Proportion of subjects with changes to QTcF from Baseline exceeding >30ms | Days 1 & 7
Proportion of subjects with changes to QTcF from Baseline exceeding >60ms | Days 1 & 7
Change in Heart Rate compared to baseline | Days 1 & 7
Change in PR Interval compared to baseline | Days 1 & 7
Change in QRS duration compared to baseline | Days 1 & 7

OTHER OUTCOMES:
Plasma concentration of MT-8554 with respect to time | Days 1 & 7
Plasma concentration of metabolite with respect to time | Days 1 & 7
Number of participants with treatment related adverse events | Days 1 to 9

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science, Study Director — Tanabe Pharma America, Inc.
Locations (1):
- Investigational center, City Name, United Kingdom